CLINICAL TRIAL: NCT05785091
Title: Correlation Between the Degree of Forward Head Posture and Hamstring Muscles Tightness in Non Specific Neck Pain
Brief Title: the Degree of Forward Head Posture and Hamstring Muscles Tightness
Status: Completed | Type: Observational
Sponsor: Holy Shaker Iskander Naroz (Other)
Responsible Party: Sponsor-Investigator, Holy Shaker Iskander Naroz, physical therapist, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 004177
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-03

CONDITIONS: Forward Head Posture
Keywords: hamstring muscles tightness; calf muscles tightness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: forward head posture with hamstring muscles tightness
- 2: forward head posture with calf muscles tightness
- 3: forward head posture and hamstring- calf muscles tightness
- 4: forward head posture and lumber inflexibility
- 5: forward head posture and hamstring- calf muscles tightness, lumber inflexibility

SUMMARY:
is the degree of forward head posture correlated with the degree of hamstring muscles tightness

DETAILED DESCRIPTION:
I will measure the degree of forward head posture by photogrammetry method and classify the degree according to its severity measuring the hamstring muscles tightness and classify it too according to its severity and calf muscle tightness lumber flexibility and correlate the to the degree of forward the forward head posture and the degree

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants 18-30 of age
2. Craniovertebral angle < 490
3. With or without neck pain

   * subjects with mechanical neck pain (in individual with chronic non-specific neck pain)
   * Subjects are not engaged in any sports or athletic routine Neck disability index >5 points

Exclusion Criteria:

.Prevalence of serious pathology (rheumatoid arthritis, ankylosing spondylitis, malignancy, infection, inflammatory disorders).

Vascular syndrome such as vertebrobasilar insufficiency Cervical spine history of trauma, fracture, congenital anomalies, or surgical intervention .

Progressive neurological deficits .

.History of lumbar and cervical herniated intervertebral disc with spinal stenosis History of neurological (Guillain-Barre, peripheral neuritis) or orthopedic disorders (osteoporosis, osteoarthritis) Moderate or severe scoliosis History of lower extremity fracture and surgery with malunion Leg length discrepancy BMI <18 or BMI >29.9

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: university students
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
correlation between the degree of forward head posture and hamstring muscles tightness in non specific neck pain | 6 month
  hamstring muscles tightness is correlated with forward head posture

SECONDARY OUTCOMES:
correlation between the degree of forward head posture and hamstring muscles tightness in non specific neck pain | 6 month
  calf muscle tightness is correlated with forward head posture

CONTACTS AND LOCATIONS:
Locations (1):
- CairoU, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
secured official researcher mail with consent form and participant approval